CLINICAL TRIAL: NCT03656588
Title: Does the Addition of Hydrogen Peroxide to Chlorhexidine Preoperative Skin Preparation Reduce the Rate of Propionibacterium Acnes Positive Culture in the Shoulder
Brief Title: Does the Addition of Hydrogen Peroxide to Chlorhexidine Skin Prep to Treat P. Acnes in the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018SNam2
Record Dates: First submitted 2018-08-23; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Propionibacterium Infection
MeSH Terms: interventions — chlorhexidine gluconate; 2-Propanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a. Standard iodine scrub, 3% hydrogen peroxide prep, follow by (Active Comparator)
  Interventions: Drug: a. Standard iodine scrub, 3% hydrogen peroxide prep, follow by ChloraPrep (2% chlorhexidine gluconate and 70% isopropyl alcohol
- b. Iodine scrub and ChloraPrep alone (Active Comparator)
  Interventions: Drug: Iodine scrub and ChloraPrep alone

INTERVENTIONS:
Drug: a. Standard iodine scrub, 3% hydrogen peroxide prep, follow by ChloraPrep (2% chlorhexidine gluconate and 70% isopropyl alcohol — a. Standard iodine scrub, 3% hydrogen peroxide prep, follow by ChloraPrep (2% chlorhexidine gluconate and 70% isopropyl alcohol
  Arms: a. Standard iodine scrub, 3% hydrogen peroxide prep, follow by
Drug: Iodine scrub and ChloraPrep alone — Iodine scrub and ChloraPrep alone
  Arms: b. Iodine scrub and ChloraPrep alone

SUMMARY:
This is a prospective, randomized controlled trial to evaluate the ability of hydrogen peroxide preparation in addition to chlorhexidine to decrease the colonization of Propionibacterium acnes(a bacteria commonly found in the dermis of the skin surrounding the shoulder in order to decrease postoperative joint infection.

ELIGIBILITY:
Inclusion Criteria:

1. All male patients (>18) undergoing shoulder arthroscopy

Exclusion Criteria:

1. Female patients
2. Patients with active acne
3. Patients who have taken antibiotics within a month of their surgery
4. Subjects allergic to any of the following agents:

   o Benzoyl peroxide
5. Subjects with psoriatic/eczematous lesions on the shoulder girdle.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
colonization of p.acnes in the dermis of the shoulder | 14 days in culture
  number of colony forming units grown in bacterial culture

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No